CLINICAL TRIAL: NCT07280390
Title: The Impact of Microplastics and Nanoplastics on Liver Health and Cardiovascular Diseases in India
Brief Title: Microplastics, Cirrhosis and Portal Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Vellore Institute of Technology University (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Additional Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: PGI/IEC/2025/EIC000779
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis; Microplastics; Portal Hypertension Related to Cirrhosis; Nanoplastics; Pollution; Cirrhosis and Chronic Liver Disease
Keywords: Microplastics; Nanoplastics; Plastic pollution; Cirrhosis; Portal hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Liver Biopsy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Cirrhosis: Cirrhosis and Portal Hypertension who are getting elective surgery or liver transplantation
  Interventions: Diagnostic Test: Assessment of microplastics in tissue

INTERVENTIONS:
Diagnostic Test: Assessment of microplastics in tissue — After meeting inclusion and exclusion criteria, 30 patients with cirrhosis will be included in this study with written informed consent from patient (surgical cases) or scheduled liver biopsy. Diagnosis of chronic liver disease will be based on history, physical examination, laboratory investigations, upper gastrointestinal endoscopy as recorded in the patient file, imaging studies (ultrasonography and doppler of splenoportal venous axis). Underlying etiology of liver disease will be recorded. Complications of cirrhosis like hepatorenal syndrome (HRS), spontaneous bacterial peritonitis (SBP), upper gastrointestinal bleed, hepatic encephalopathy, acute kidney injury will be recorded from the patient's casefile.
  Tissue Sample Processing Standard laboratory solvents (i.e., acetonitrile, methanol, and water (LiChrosolv and SupraSolv grade) will be procured. The contact of laboratory surfaces and equipment will be minimized to reduce the risk of background contamination by plastics.

SUMMARY:
Cirrhosis and portal hypertension are associated with an hyperdynamic circulation and hepatic inflammation, leading to complications like ascites, variceal bleeding, acute kidney injury, and higher infection risk. Microplastics (MPs) are a global plastic pollution issue, and studies have found plastic MPs or nanoparticles (NPs) contaminating human, animal and environmental ecosystems.It has been noted that the accumulation of MPs increases with a reduction in size of the plastic particle. MPs are categorized into primary particles such as manufactured plastics including pellets and cosmetic microbeads and secondary particles which originate from mechanical and ultraviolet disruption of large plastic particles. MPs can be ingested via food or beverages, especially plastic packaged comestibles or inhaled as environmental pollutants. Contamination of medications such as antibiotics, intravenous fluids, albumin and medical devices is another source of exposure to microplastics in patients with chronic liver disease (CLD)In particular exposure to endoscopic interventions, liver biopsy, and invasive procedures such as paracentesis and interventional radiology procedures can lead to plastic exposure and deposition of MPs in the liver and other tissues in patients with cirrhosis. It may be hypothesized that these may contribute to hepatic inflammation and progression of cirrhosis and portal hypertension.

Globally, there is new research on the influence of MPs on the environment, plant and animal ecosystems and human health.

Polystyrene (PS) microspheres that concentrate in the liver, intestine and the kidneys of mammals disrupt lipid and energy metabolism, impair mucus secretion, and alter the microbiome. Therefore, studies are required to assess how and to what extent, MPs impact human health, and affect chronic diseases like cirrhosis and reduce longevity.

In the proposed study we will assess the presence of MPs in the liver, kidneys and intestine of patients with liver cirrhosis and compare it with those without underlying liver disease and determine the impact on portal hypertension and fibrosis, and cardiovascular and metabolic function.

DETAILED DESCRIPTION:
First, because the methodology requires chemical digestion, it is unclear where in the liver MPs are deposited. For instance, it is indeterminate if MPs are deposited intracellularly, in Kupffer cells, endothelium or hepatocytes/cholangiocytes. In the present study we intend to perform histopathological assessments of the liver tissue to determine the presence of the MPs.

* Furthermore, our study will assess various polymer types of MP in cirrhotic liver tissue including commonly observed plastic polymers PS (polystyrene), PE (polyethylene), PP (polypropylene), PVC (polyvinyl chloride), PET (polyethylene terephthalate), PC (polycarbonate), and PMMA (polymethyl methacrylate).
* Therefore, we need to assess potential cellular sites of deposition in the liver. If the MPs were in the systemic circulation, without any liver parenchymal residues, such particles should also be identified in spleen and kidney samples.
* In the present study we intend to overcome these limitations by histopathology and electron microscopy of the liver tissue which should clarify the specific accumulation sites.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-70 years
* Cirrhosis, as diagnosed by histology or clinical, laboratory and USG findings.
* Undergoing elective surgery or liver transplantation

Exclusion Criteria:

* • Hepatocellular carcinoma

  * Pregnancy or lactation
  * Patients with HIV or retroviral therapy
  * Prior liver interventions like locoregional therapy, presence of HCC, prior abdominal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis Healthy liver control tissue will be taken from autopsy patients with consent
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to assess MPs in human liver tissue, analysing their morphology, size, and composition (4-30 µm). We will examine tissue samples from the liver inpatients with cirrhosis as compared with controls without cirrhosis | At time of enrolment
  MPs in liver cirrhosis

SECONDARY OUTCOMES:
• Identification of Various polymer types, including PS, PVC, PET, PMMA, POM, and PP and surface alterations indicative of long-term deposition. | At enrolment
  Assessment of type of microparticles
• Determination of plastic pollution exposure in patients with cirrhosis by detailed history of diet, oral and parenteral medication, interventions including prior biopsy and endoscopy | At the time of elective endoscopy
  Assessment of gastric and duodenal mucosa for micronanoplastics during elective endoscopy.
Assessment of micronanoplastics in peripheral blood | At enrolment
  Dried blood spots assessment of micronanoplastics

OTHER OUTCOMES:
Association of microplastics with degree of liver fibrosis and inflammation | At enrolment
  Comparison of presence of microplastics with histopathological inflammation and presence of fibrosis grade.

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, Principal Investigator — PGIMER Chandigarh
Locations (1):
- PGIMER Chandigarh, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided